CLINICAL TRIAL: NCT00662831
Title: A 6 Month, Prospective, Randomized, Double Blind, Placebo-Controlled, Parallel Group, Multiple Center Trial To Evaluate The Efficacy And Safety Of Fragmin In The Treatment Of Chronic Neuroischaemic Foot Ulcers In Diabetic Patients
Brief Title: Study Of The Effect Of Fragmin In The Treatment Of Neuroischaemic Foot Ulcers In Diabetic Patients
Acronym: FEENICS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6301083
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcers Neuroischaemic
MeSH Terms: conditions — Diabetic Foot | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Active study treatment
  Interventions: Drug: Fragmin/ Dalteparin Sodium
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo for Fragmin/ Dalteparin Sodium

INTERVENTIONS:
Drug: Fragmin/ Dalteparin Sodium — Pre-filled syringes containing a single dose of 5000 IU Fragmin/ Dalteparin Sodium.
  Arms: Active
Drug: Placebo for Fragmin/ Dalteparin Sodium — Pre-filled syringes containing a single dose of placebo for 5000 IU Fragmin/ Dalteparin Sodium.
  Arms: Placebo

SUMMARY:
The purpose of the study isto see the effect of Fragmin on the healing of diabetic foot ulcers by determining the number of subjects with ≥50% reduction in ulcer surface area including intact skin healing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age with type 1 or type 2 diabetes.
* Subjects with peripheral occlusive arterial disease (PAOD) and a neuropathy disability score (NDS) of >3

Exclusion Criteria:

* Subjects who have undergone vascular reconstruction or angioplasty less than 1 month prior to randomization. Subjects with an ulcer grading of 0 or 3 and staging of A, B or D according to the University of Texas wound classification system.
* Subjects with a known bleeding disorder or evidence of active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- Austria (2):
  - Pfizer Investigational Site, Klagenfurt
  - Pfizer Investigational Site, Vienna
- Pfizer Investigational Site, Ransart, Belgium
- Canada (2):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Montreal, Quebec
- Czechia (2):
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Zlín
- Denmark (6):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Hvidovre
  - Pfizer Investigational Site, Koebenhavn NV
  - Pfizer Investigational Site, Odense C
  - Pfizer Investigational Site, Sønderborg
- Pfizer Investigational Site, Tampere, Finland
- Pfizer Investigational Site, Karlsbad, Germany
- Greece (3):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Melissia/Athens
  - Pfizer Investigational Site, Thessaloniki
- Italy (4):
  - Pfizer Investigational Site, San Giovanni Rotondo, FG
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Roma
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Pfizer Investigational Site, Tønsberg, Norway
- Poland (5):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Puławy
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Spain (3):
  - Pfizer Investigational Site, Getafe, Madrid
  - Pfizer Investigational Site, Girona
  - Pfizer Investigational Site, Madrid
- Sweden (3):
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
- Ukraine (4):
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Odesa
- United Kingdom (8):
  - Pfizer Investigational Site, Barnsley
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Colchester
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Ipswich
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Peterborough

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301083&StudyName=Study%20Of%20The%20Effect%20Of%20Fragmin%20In%20The%20Treatment%20Of%20Neuroischaemic%20Foot%20Ulcers%20In%20Diabetic%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalteparin: Dalteparin 5000 International Units (IU) (0.2 milliliter [mL]) subcutaneously (s.c.) once daily for 24 weeks or early termination (ET).
- Placebo: Placebo (0.2 mL normal saline) administered s.c. once daily for 24 weeks or ET.
Period: Overall Study
Arm/Group | Dalteparin | Placebo
Started | 184 | 92
Completed | 78 | 33
Not Completed | 106 | 59
Not completed — Death | 4 | 1
Not completed — Lack of Efficacy | 6 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 62 | 31
Not completed — Protocol Violation | 8 | 4
Not completed — Adverse Event | 23 | 16

BASELINE CHARACTERISTICS:
Groups:
- Dalteparin: Dalteparin 5000 International Units (IU) (0.2 mL) subcutaneously (s.c.) once daily for 24 weeks or early termination (ET).
- Total: Total of all reporting groups
Arm/Group | Dalteparin | Placebo | Total
Number analyzed (Participants) | 184 | 92 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.3) | 64.7 (10.9) | 64.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 30 | 93
  Male | 121 | 62 | 183

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Greater Than or Equal to 50 Percent Reduction in Ulcer Surface Area Including Intact Skin Healing
Description: University of Texas (UT) system assesses ulcer depth, wound infection and clinical signs of lower-extremity ischemia. UT Wound Classification (1C/2C) was based on grade (0= healed site to 3= penetrating wound to bone or joint) and stage (A= clean wounds to D= ischaemic infected wounds) of wounds. Participants were evaluated at 4 stratums: Stratum 1: Toe pressure>30 mm of mercury (mmHg) and UT grade and stage 1C. Stratum 2: Toe pressure<=30 mmHg and UT grade and stage 1C. Stratum 3: Toe pressure>30 mmHg and UT grade and stage 2C. Stratum 4: Toe pressure<=30 mmHg and UT grade and stage 2C.
Time Frame: Week 24 [end of treatment (EOT)] or early termination
Population: Intention to treat (ITT) population included all participants who were randomized. Last observation carried forward (LOCF) method was used. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Number; unit: participants
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
participants
  Stratum 1 (n= 97, 49) | 68 | 31
  Stratum 2 (n= 39, 19) | 23 | 14
  Stratum 3 (n= 29, 14) | 21 | 10
  Stratum 4 (n= 19, 10) | 9 | 6

2. Secondary Outcome: Number of Participants With Intact Skin Healing
Description: Intact skin healing was defined as 100 percent reduction in ulcer surface area with full epithelialisation. UT system assesses ulcer depth, wound infection and clinical signs of lower-extremity ischemia. Participants were evaluated at 4 stratums: Stratum 1: Toe pressure>30 mm of mercury (mmHg) and UT grade and stage 1C. Stratum 2: Toe pressure<=30 mmHg and UT grade and stage 1C. Stratum 3: Toe pressure>30 mmHg and UT grade and stage 2C. Stratum 4: Toe pressure<=30 mmHg and UT grade and stage 2C.
Time Frame: Week 24 (EOT) or early termination
Population: ITT population included all participants who were randomized. LOCF method was used. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Number; unit: participants
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
participants
  Stratum 1 (n= 97, 49) | 35 | 16
  Stratum 2 (n= 39, 19) | 15 | 4
  Stratum 3 (n= 29, 14) | 8 | 4
  Stratum 4 (n= 19, 10) | 1 | 4

3. Secondary Outcome: Number of Participants Who Underwent Any Amputation
Description: Any amputation included both major and minor amputations. A major amputation was defined as above the ankle and was reported as below-the-knee and above-the-knee amputations. A minor amputation was defined as below the ankle amputation.
Time Frame: Week 24 (EOT) or early termination
Population: ITT population included all participants who were randomized.
Measure: Number; unit: participants
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 180 | 90
participants | 8 | 2

4. Secondary Outcome: Number of Participants Who Underwent Major and Minor Amputation
Description: A major amputation was defined as above the ankle and was reported as below-the-knee and above-the-knee amputations. A minor amputation was defined as below the ankle amputation.
Time Frame: Week 24 (EOT) or early termination
Population: ITT population included all participants who were randomized.
Measure: Number; unit: participants
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 180 | 90
participants
  Major amputation | 2 | 1
  Minor amputation | 7 | 1

5. Secondary Outcome: Number of Participants With Greater Than or Equal to 50 Percent Reduction in Ulcer Surface Area Excluding Intact Skin Healing
Description: as for outcome 1
Time Frame: Week 24 (EOT) or early termination
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
participants
  Stratum 1 (n= 97, 49) | 33 | 15
  Stratum 2 (n= 39, 19) | 8 | 10
  Stratum 3 (n= 29, 14) | 13 | 6
  Stratum 4 (n= 19, 10) | 8 | 2

6. Secondary Outcome: Number of Participants Who Died
Time Frame: Week 24 (EOT) or early termination
Population: ITT population included all participants who were randomized.
Measure: Number; unit: participants
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
participants | 4 | 3

7. Secondary Outcome: Number of Participants With Major Cardiovascular Disease Events (MCVE)
Description: Major cardiovascular events were defined as death due to vascular cause; non-fatal myocardial infarction (MI) excluding procedure related to MI; coronary revascularization procedures not related to MIs; hospitalization for unstable angina or non-fatal stroke.
Time Frame: Week 24 (EOT) or early termination
Population: The data was not analyzed as planned because the study enrollment was terminated before the planned number of randomized participants was obtained.
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Intact Skin Healing
Description: Median time taken to achieve intact skin healing which was defined as 100 percent reduction in ulcer surface area with full epithelialisation.
Time Frame: Week 24 (EOT) or early termination
Population: as for outcome 7
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Median Time to First Amputation
Time Frame: Week 24 (EOT) or early termination
Population: as for outcome 7
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D)- Utility Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. It assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline and Week 24 (EOT or early termination)
Population: ITT population included all participants who were randomized. Participants were only considered when all items contributing to the score had been answered. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 182 | 88
Units on a scale
  Baseline | 0.60 (0.26) | 0.60 (0.30)
  EOT (n= 154, 74) | 0.70 (0.22) | 0.60 (0.33)

11. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline and Week 24 (EOT or early termination)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 182 | 91
mm
  Baseline | 60.20 (18.68) | 55.30 (19.72)
  EOT (n= 157, 76) | 63.30 (18.76) | 60.70 (18.02)

12. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) Score
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline and Week 24 (EOT or early termination)
Population: ITT population included all participants who were randomized. This was calculated only when more than half of the questions within dimension were answered. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 90
Units on a scale
  Baseline: Physical Functioning | 34.70 (12.06) | 32.50 (10.96)
  Baseline: Role-Physical | 35.40 (11.22) | 35.20 (11.41)
  Baseline: Bodily Pain | 42.30 (11.19) | 40.30 (11.52)
  Baseline: General Health | 42.30 (5.52) | 42.60 (5.10)
  Baseline: Visibility | 48.30 (5.63) | 48.70 (5.02)
  Baseline: Social Functioning | 33.00 (6.49) | 33.10 (6.90)
  Baseline: Role-Emotional | 39.10 (13.48) | 38.30 (13.49)
  Baseline: Mental Health | 41.90 (6.57) | 41.30 (6.72)
  Baseline: Physical (PCS) | 38.10 (9.42) | 36.70 (8.75)
  Baseline: Mental (MCS) | 42.40 (7.26) | 42.80 (7.37)
  EOT: Physical Functioning (n= 156, 76) | 37.10 (11.71) | 35.50 (11.39)
  EOT: Role-Physical (n= 155, 76) | 39.30 (11.25) | 37.50 (11.31)
  EOT: Bodily Pain (n= 156, 76) | 47.50 (10.30) | 45.00 (10.73)
  EOT: General Health (n= 156, 76) | 42.50 (5.10) | 42.80 (5.15)
  EOT: Visibility (n= 156, 76) | 48.20 (5.58) | 48.80 (5.15)
  EOT: Social Functioning (n= 152, 73) | 33.30 (6.13) | 32.30 (5.83)
  EOT: Role-Emotional (n= 155, 76) | 41.20 (13.44) | 38.80 (13.48)
  EOT: Mental Health (n= 156, 76) | 41.90 (6.20) | 42.00 (6.80)
  EOT: Physical (PCS) (n= 151, 73) | 41.70 (9.04) | 40.10 (8.60)
  EOT: Mental (MCS) (n= 151, 73) | 42.10 (6.89) | 41.60 (6.46)

13. Secondary Outcome: 11-point Likert Pain Scale
Description: The 11 point Likert pain scale which used a 0 (no pain) to 10 (worst possible pain) point rating system was used to assess participant's pain score. No distinction was made between neuropathy and inflammatory (nociceptive) pain.
Time Frame: Baseline and Week 24 (EOT or early termination)
Population: ITT population included all participants who were randomized. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 183 | 89
Units on a scale
  Baseline | 4.20 (2.76) | 4.50 (2.83)
  EOT (n= 155, 75) | 2.10 (2.27) | 2.50 (2.54)

14. Secondary Outcome: Transcutaneous Local Tissue Oxygenation (pO2)
Description: Transcutaneous pO2 was assessed at the dorsum of the foot in the first intermetatarsal space using an appropriately calibrated instrument. The skin oxygen partial pressure was determined by measuring the oxygen reduction current by means of a measuring cell.
Time Frame: Baseline and Week 24 (EOT or early termination)
Population: ITT population included all participants who were randomized. Participants were analyzed at selected sites only, based on availability. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 47 | 26
Units on a scale
  Baseline | 31.80 (21.29) | 36.00 (17.11)
  EOT (n= 32, 19) | 38.80 (19.58) | 39.70 (16.18)

15. Other Pre Specified Outcome: Number of All Hemorrhages
Description: Major hemorrhages: defined as fatal bleeding, clinically overt bleeding causing a fall in hemoglobin more than or equal to 20 gram (g)/litre (L) (2 g/ decilitre [dL]), clinically overt bleeding leading to transfusion of more than or equal to 2 units of whole blood or red cells, or symptomatic bleeding in areas of special concern (intracranial, retroperitoneal, intraocular, intraspinal, pericardial, intramuscular with compartmental syndrome, or intraarticular). Minor hemorrhages: defined as bleeding that did not meet the definition of major bleeding.
Time Frame: Week 24 (EOT) or early termination
Population: Safety analysis population included all participants who were known to have taken at least one dose of the study medication.
Measure: Number; unit: hemorrhages
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
hemorrhages | 10 | 2

16. Other Pre Specified Outcome: Number of Major and Minor Hemorrhages
Description: as for outcome 15
Time Frame: Week 24 (EOT) or early termination
Population: as for outcome 15
Measure: Number; unit: hemorrhages
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
hemorrhages
  Major hemorrhages | 2 | 0
  Minor hemorrhages | 8 | 2

17. Other Pre Specified Outcome: Number of Clinically Relevant Minor Hemorrhages and Trivial Hemorrhages
Description: Clinically relevant minor (non-major) bleeding was defined as any bleeding compromising hemodynamics, leading to hospitalization, subcutaneous haematoma more than 25 cm^2, intramuscular haematoma, epistaxis lasting for more than 5 minutes, spontaneous gingival bleeding, macroscopic hematuria and gastrointestinal hemorrhage (including at least 1 episode of melaena or hematemesis), rectal blood loss, hemoptysis, and any other bleeding with clinical consequences. Trivial bleeding was defined as all minor bleeding that did not meet the definition of clinically relevant minor bleeding.
Time Frame: Week 24 (EOT) or early termination
Population: as for outcome 15
Measure: Number; unit: hemorrhages
Arm/Group | Dalteparin | Placebo
Number analyzed (Participants) | 184 | 92
hemorrhages
  Clinically relevant minor hemorrhages | 5 | 1
  Trivial hemorrhages | 3 | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dalteparin | Placebo
Serious Adverse Events (participants affected / at risk) | 33/184 | 18/92
Other Adverse Events (participants affected / at risk) | 76/184 | 36/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=184) | Placebo (N=92)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Condition aggravated (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Ulcer (General disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Arteriosclerotic gangrene (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 1
Erysipelas (Infections and infestations) | 1 | 3
Gangrene (Infections and infestations) | 4 | 0
Infected skin ulcer (Infections and infestations) | 3 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 2
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Strangury (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin (N=184) | Placebo (N=92)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Monocytopenia (Blood and lymphatic system disorders) | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 1
Injection site haematoma (General disorders) | 7 | 0
Injection site pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 3
Pain (General disorders) | 1 | 1
Ulcer (General disorders) | 3 | 4
Liver disorder (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Diabetic foot infection (Infections and infestations) | 4 | 2
Erysipelas (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 6 | 5
Infection (Infections and infestations) | 4 | 0
Influenza (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 3 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Antibiotic resistant Staphylococcus test positive (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose abnormal (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 | 3
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study enrollment was terminated before planned number of participants was obtained. Although randomized participants were allowed to complete entire course of therapy according to protocol and study status was therefore designated as completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.